CLINICAL TRIAL: NCT04257045
Title: Factors Influencing Cascade Testing Among Women With Hereditary Gynecological Cancers and Their Relatives
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019-0239; NCI-2019-05371 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0239 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-02-04; First posted 2020-02-05 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Breast Carcinoma; Deleterious CDH1 Gene Mutation; Deleterious DICER1 Gene Mutation; Deleterious SMARCA4 Gene Mutation; Deleterious STK11 Gene Mutation; Endometrial Carcinoma; Fallopian Tube Carcinoma; Ovarian Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (interview, survey): STEP I: Patients and first degree relatives participate in semi-structure, in-depth interviews about genetic testing over 45-60 minutes.
  STEP II: Patients and first degree relatives complete survey questionnaires over 20 minutes.
  Interventions: Other: Interview; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Interview — Participate in semi-structure, in-depth qualitative interviews
Other: Questionnaire Administration — Complete questionnaires
Other: Survey Administration — Complete survey

SUMMARY:
This trial collects information about factors that affect communication of genetic test results, decision-making, and access to genetic testing in women with hereditary gynecological cancers. Studying individuals who are positive for a genetic mutation and immediate biological family members (including a parent, full-sibling, or child) may help identify cancer genes and other persons at risk.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify and explore factors influencing the communication of genetic testing results from probands (patients with confirmed hereditary cancer predisposition syndrome) to their first-degree relatives. (Step 1) II. Identify and explore factors influencing decision making and pursuit of cascade testing among first-degree relatives of probands. (Step 1) III. Estimate the uptake of cascade testing by first-degree relatives of probands at a safety-net hospital and the uptake of cascade testing by first-degree relatives of probands at a comprehensive cancer center. (Step 2) IV. Estimate the frequency of reported factors that influence communication, decision-making, and pursuit of cascade testing among probands and their first-degree family members at a safety-net hospital and at a comprehensive cancer center. (Step 2) V. Explore similarities and differences in cascade genetic testing rates and reported barriers to cascade genetic testing of first-degree relatives at probands from a safety-net hospital and a comprehensive cancer center. (Step 2)

OUTLINE:

STEP I: Patients and first degree relatives participate in semi-structure, in-depth interviews about genetic testing over 45-60 minutes.

STEP II: Patients and first degree relatives complete survey questionnaires over 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 (PROBANDS): Speaks and/or reads English or Spanish
* STEP 1 (PROBANDS): Currently receiving diagnostic, treatment, or follow-up care in the outpatient gynecologic oncology and medical oncology clinics at LBJ
* STEP 1 (PROBANDS): Has completed genetic counseling, with pedigree available in the medical record (LBJ)
* STEP 1 (PROBANDS): Diagnosed with female-breast, ovarian, fallopian tube, primary peritoneal, endometrial cancer on or after January 1, 2014
* STEP 1 (PROBANDS): Has a confirmed deleterious or suspected deleterious (pathogenic) variant in a hereditary gynecologic or breast cancer predisposition gene (including BRCA1, BRCA2, MLH1, MSH2, MSH6, PMS2, EPCAM, BRIP1, PALB2, RAD51C, RAD51D, STK11, DICER1, SMARCA4, ATM, CHEK2, PTEN, TP53, CDH1, BARD1)
* STEP 1 (FIRST-DEGREE RELATIVE [FDR]): Speaks and/or reads English or Spanish
* STEP 1 (FDR): Is a first-degree relative of proband (son, daughter, full-brother, full-sister, mother, father)
* STEP 1 (FDR): Is present with proband at time of recruitment, or can be contacted by telephone via a United States (U.S.) telephone number
* STEP 1 (FDR): Is aware of proband's genetic testing result/mutation status, per proband report
* STEP 2 (PROBANDS): Speaks or reads English or Spanish
* STEP 2 (PROBANDS): Currently receives diagnostic, treatment, or follow-up care for female-breast cancer in the outpatient medical oncology clinics at LBJ; or currently receives diagnostic, treatment, or follow-up care for ovarian, fallopian tube, primary peritoneal or endometrial cancer in the outpatient gynecologic oncology clinic at LBJ or the outpatient gynecologic oncology clinic at The University of Texas MD Anderson Cancer Center (MD Anderson)
* STEP 2 (PROBANDS): Diagnosed with eligible cancer on or after January 1, 2014
* STEP 2 (PROBANDS): Has completed genetic counseling, with a pedigree available in the medical record (LBJ) or internal clinical and research database (progeny at MD Anderson)
* STEP 2 (PROBANDS): Has a confirmed deleterious or suspected deleterious (pathogenic) variant in a hereditary gynecologic or breast cancer predisposition gene (including BRCA1, BRCA2, MLH1, MSH2, MSH6, PMS2, EPCAM, BRIP1, PALB2, RAD51C, RAD51D, STK11, DICER1, SMARCA4, ATM, CHEK2, PTEN, TP53, CDH1, BARD1)
* STEP 2 (FDR): Speak and/or reads English or Spanish
* STEP 2 (FDR): First-degree relative of proband (son, daughter, full-brother, full-sister, mother, father)
* STEP 2 (FDR): Is present with proband at time of recruitment, or can be contacted by telephone via a U.S. telephone number
* STEP 2 (FDR): Is aware of proband's genetic testing result/mutation status, per proband report

Exclusion Criteria:

* STEP 1 (PROBANDS): No longer receives outpatient care at LBJ
* STEP 1 (PROBANDS): Has a negative genetic testing result, a result identifying only a variant of uncertain significance, or results and pedigree that cannot be confirmed in the electronic medical record
* STEP 1 (PROBANDS): Is unwilling or unable to provide informed consent
* STEP 1 (FIRST-DEGREE RELATIVE [FDR]): Unwilling or unable to provide informed consent
* STEP 2 (PROBANDS): No longer receives outpatient care at LBJ or MD Anderson
* STEP 2 (PROBANDS): Has a negative genetic testing result, a result identifying only a variant of uncertain significance, or results and pedigree that cannot be confirmed in the electronic medical record
* STEP 2 (PROBANDS): Unwilling or unable to provide informed consent
* STEP 2 (PROBANDS): Participated in step 1 interviews
* STEP 2 (FDR): Unwilling or unable to provide informed consent
* STEP 2 (FDR): Reports no knowledge of proband's genetic testing status
* STEP 2 (FDR): Participated in step 1 interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients currently receiving diagnostic, treatment, or follow-up care in the outpatient Gynecologic Oncology and Medical Oncology clinics at Lyndon B. Johnson Hospital (LBJ), and their first-degree relatives.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Factors influencing decision-making and communication of genetic test results (Step 1) | Up to 3 years
Rates of cascade testing among first-degree relatives (Step 2) | Up to 3 years
  Will be calculated using summary statistics. Will construct a generalized linear mixed model (GLMM) with a logit link function to estimate rate of cascade testing among first-degree relatives.
Genetic testing rate (Step 2) | Up to 3 years
  Will construct a model with no predictors and will calculate the probability of genetic testing using the model's intercept as well as calculate the 95% confidence interval of this probability. Will then test factors associated with testing rates (including site [Lyndon B. Johnson Hospital (LBJ) vs. MD Anderson (MDA)], socioeconomic, demographic, medical history, and determinants) by including these as independent variables in our GLMMs.
Frequency of reported barriers (Step 2) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Rauh-Hain, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org